CLINICAL TRIAL: NCT04515290
Title: A Phase IIa Clinical Trial on TSG-01 in the Treatment of Chronic Heart Failure in Patients With Coronary Heart Disease.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Hongyitang Biopharmaceutical Technology Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HYT-CT-01
Record Dates: First submitted 2020-08-13; First posted 2020-08-17 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Chronic Heart Failure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TSG-01-H (Experimental): Two tablets of TSG-01 per time.
  Interventions: Drug: TSG-01
- TSG-01-L (Experimental): One tablet of TSG-01 and One tablet of Placebo per time.
  Interventions: Drug: TSG-01 and Placebo
- Control (Placebo Comparator): Two tablets of Placebo per time.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TSG-01 — Two tablets of TSG-01 (0.35g/tablet) were given by oral with 3 times a day for 12 weeks; High dose group.
  Arms: TSG-01-H
Drug: TSG-01 and Placebo — One tablet of TSG-01 (0.35g/tablet) and one tablet of placebo (0.35g/tablet) were given by oral with 3 times a day for 12 weeks; Low dose group.
  Arms: TSG-01-L
Drug: Placebo — Two tablets of placebo (0.35g/tablet) were given by oral with 3 times a day for 12 weeks.
  Arms: Control

SUMMARY:
The purpose of this study is to assess the safety, efficacy and optimal dose of TSG-01, an innovative drug with ginsenosides as its main components, in the treatment of patients with chronic heart failure(CHF). Preclinical studies have revealed that TSG-01 promote myocardial energy metabolism and ATP production, reduce the damage of human pulmonary microvascular endothelial cell connection, resist arrhythmia, and regulate the lipid metabolism disorder caused by myocardial ischemia. Results from CHF animal models(dog, rat) showed that TSG-01 significantly increase coronary blood supply, improve myocardial contractility, reduce heart expansion and pulmonary edema. Besides its potency of improving heart function, TSG-01 was found to induce diuresis without obvious effect on urine potassium in rats. TSG-01 has been approved by CFDA for a clinical trial on the treatment of CHF (Approval No. 2018L03012). A randomized, double-blind, multicenter, placebo-controlled phase IIa clinical trial is now being conducted in 5 hospitals in China. A total of 90 cases of CHF caused by coronary heart disease are included and randomly divided into three groups: high-dose, low-dose of TSG-01 and placebo group. NYHA functional class, 6-minute walk test(6MHWT) distance, NT-proBNP, left ventricular ejection fraction(LVEF), echocardiographic parameters (LVESV, LVEDV, and heart size) and MLHFQ score are measured before, during and after treatment to evaluate the benefits of TSG-01 therapy in patients with CHF.

ELIGIBILITY:
Inclusion Criteria:

* Age: 40 to 75 years.
* Have chronic heart failure(CHF) due to ischemic causes and defined as NYHA classification of III.
* Left ventricular ejection fraction (LVEF) of ≤45% and ≥25% as determined by improved biplane Simpson method
* NT-proBNP≥450pg/ml
* Be on a stable regime of standardized therapy for CHF at least 2 weeks prior to receiving study medication and are respected to remain on a stable regime throughout the duration of the trial without the need to receive intravenously vasoactive agents or/and diuretics. Standardized therapy includes ACEI/ARB, beta-blocker, aldosterone receptor antagonist, diuretic, digitalis.
* Is able to understand the trial and provide informed consent.

Exclusion Criteria:

* Has hypertensive cardiopathy, pulmonary heart disease, congenital heart disease, moderate to severe pulmonary hypertension (pulmonary artery pressure ≥ 40mmHg), moderate to severe cardiac valve stenosis or insufficiency, any type of cardiomyopathy(hypertrophic, restrictive or dilated cardiomyopathy); moderate to severe pericardial effusion, constrictive pericarditis, and heart failure caused by arrhythmia.
* Has noncardiogenic heart failure caused by diseases in kidney, lung, liver, or by rheumatic immune disorders, severe infection and chemical factors (chemotherapy, alcohol, etc.).
* Has active tuberculosis or systemic lupus erythematosus (SLE)
* Had acute myocardial infarction, biventricular pacemaker implantation for cardiac resynchronization, cardiothoracic surgery or was complicated with acute coronary syndrome, pulmonary embolism and acute cerebrovascular disease within 3 months prior to receiving study medication.
* Had symptomatic ventricular tachycardia or pleomorphic ventricular tachycardia, cardiogenic shock (CGS), a progressive exacerbation of unstable angina, uncontrolled malignant arrhythmia, second degree sinoatrial or AV block Mobitz Type II or above without pacemaker implantation, QTc>550 ms and heart rate <50 bmp. Had uncontrolled hypertension, systolic blood pressure≥180/mmHg and/or diastolic blood pressure≥110mmHg, or hypotension with systolic blood pressure<90mmHg and/or diastolic blood pressure<60mmHg.
* Had coronary revascularization procedure (percutaneous or surgical) within 12 weeks prior to receiving study medication or be expected to have coronary revascularization or left ventricular remodeling operation in next 12 weeks.
* Has hepatic abnormality defined as ALT≥1.5 times the upper limit of normal, or has impaired renal function with Cr≥1.5 times the upper limit of normal. Has severe anemia (Hb<70g/L), pheochromocytoma, hematopathy, gastrointestinal bleeding (consecutive fecal occult blood tests positive, except bleeding caused by hemorrhoids or other anal diseases).
* Has a body weight>200kg.
* The subject has the need for mechanical ventilation, or has a history of a stroke or any malignancy within 4 weeks prior to receiving study medication.
* Has psychosis with poor control, or is a drug addict who has not been detoxified.
* Allergic to the study drug.
* Has participated in any clinical trial involving experimental therapy 3 months prior to screening.
* If female, being pregnant or lactating, or plan to get pregnant in next 3 months.
* Has a survival time less than 3 months according to the investigator's judgement.
* Subject who are taking Entresto (Sacubitril Valsartan Sodium Tablets) medication.
* Unable to complete the study or comply with the requirements of the study (for management or other reasons) according to the investigator's judgement.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2020-05-07 (Actual); Primary Completion 2022-04-22 (Actual); Study Completion 2022-04-22 (Actual)

PRIMARY OUTCOMES:
New York Heart Association (NYHA) Classification | 12th week after intervention
  Change from baseline and placebo in NYHA class status. NYHA Classification is a heart function classification which divides impaired cardiac function into four levels according to the action capacity of the patient. And among NYHA classification, Class I represents the mildest symptoms, while Class IV represents the most severe case.
Six(6)-minute walk test | 12th week after intervention
  To measure the distance that the patient is instructed to walk along a hallway as far as he(or she) can in 6 minutes.

SECONDARY OUTCOMES:
Change of NT-proBNP (N-Terminal Pro-B-Type Natriuretic Peptide) Level from baseline and placebo | 12th week after intervention
Change in LVEF from screening/baseline as determined by echocardiography | 12th week after intervention
Change in LVESV from screening/baseline as determined by echocardiography | 12th week after intervention
Change in LVEDV from screening/baseline as determined by echocardiography | 12th week after intervention
Change in cardiac size from screening/baseline as determined by echocardiography | 12th week after intervention
Minnesota Living with Heart Failure Questionnaire (MLHFQ) | 12th week after intervention

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Henan Province Hospital of TCM, Zhengzhou, Henan
  - The first Affiliated Hospital of Henan University of CM, Zhengzhou, Henan
  - Affiliated Hospital of Nanjing University of Chinese Medicine, Nanjing, Jiangsu
  - Shanghai Shuguang Hospital, Shanghai, Shanghai Municipality
  - Zhejiang Provincial Hospital of Chinese Medicine, Hangzhou, Zhejiang